CLINICAL TRIAL: NCT02587351
Title: Beta-Blockers for the Prevention of Acute Exacerbations of COPD
Brief Title: Beta-Blockers for the Prevention of Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: University of Minnesota (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1512M81981
Record Dates: First submitted 2015-10-19; First posted 2015-10-27 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Exacerbation; Lung function; Cardiac; Cardiovascular; Beta blockers; Metoprolol succinate; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoprolol succinate (Active Comparator): Metoprolol succinate extended release tablets (50 mg) starting dose followed by a dose titration procedure which will result in a final dose of 25mg (1/2 of one tablet daily), 50 mg, or 100 mg (two tablets daily).
  Interventions: Drug: Metoprolol succinate
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metoprolol succinate — Extended release Metoprolol succinate
  Other Names: Metoprolol Succinate ER; Toprol XL
  Arms: Metoprolol succinate
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, prospective, randomized, double-blind, placebo-controlled trial that will enroll 1028 patients with at least moderately severe COPD over a three year period and follow them at regular intervals for one year. The primary endpoint is time to first acute exacerbation. Secondary endpoints include rates and severity of COPD exacerbations, cardiovascular events, all-cause mortality, lung function, dyspnea, quality of life and metoprolol-related side effects.

DETAILED DESCRIPTION:
Hypothesis The primary hypothesis is that metoprolol succinate will reduce the risk of COPD exacerbations as compared to placebo. The secondary hypothesis is that metoprolol succinate will not adversely impact lung function, exercise tolerance, dyspnea or quality of life as compared to placebo.

Study Flow Patients will be screened and then randomized over a 2 week period and will then undergo a dose titration period for the following six weeks. Thereafter patients will be followed for 42 additional weeks on their target dose of metoprolol or placebo followed by a 4 week washout period.

Specific Aims:

Primary: To determine the effect of once daily metoprolol succinate compared with placebo on the time to first exacerbation in moderate to severe COPD patients who are prone to exacerbations and who do not have absolute indications for beta-blocker therapy.

Secondary: To estimate the effect of metoprolol succinate compared with placebo on:

1. The rate and severity of COPD exacerbations over 12 months
2. Incidence and severity of metoprolol-related side effects including those that require cessation of drug
3. Lung function as assessed by spirometry, dyspnea as assessed by the Modified Medical Research Council Scale (MMRC) and San Diego Shortness of Breath Questionnaire, exercise tolerance as measured by six minute walk test (6MWD), and quality of life as assessed by the Short Form 36, St. Georges Respiratory Questionnaire (SGRQ) and COPD Assessment Test (CAT) and Personal HEART Score.
4. Hospitalizations
5. The rate of major adverse cardiovascular events (MACE) (defined by cardiovascular death, hospitalization for myocardial infarction, heart failure, or stroke), percutaneous coronary intervention or coronary artery bypass grafting
6. All-cause mortality

Secondary subgroup analyses for 1) cardiovascular risk based on Personal HEART Score and 2) age greater versus less than 65.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ≥ 40 and less than 85 years of age
2. Clinical diagnosis of at least moderate COPD as defined by the Global Initiative for Obstructive Lung Disease (GOLD) criteria (53):

   * Post bronchodilator FEV1/FVC < 70% (Forced expiratory volume in 1 second/ forced vital capacity),
   * Post bronchodilator FEV1 < 80% predicted, with or without chronic symptoms (i.e., cough, sputum production).
3. Cigarette consumption of 10 pack-years or more. Patients may or may not be active smokers.
4. To enrich the population for patients who are more likely to have acute exacerbations (54), each subject must meet one or more of the following 4 conditions:

   * Have a history of receiving a course of systemic corticosteroids and/or antibiotics for respiratory problems in the past year,
   * Visiting an Emergency Department for a COPD exacerbation within the past year, or
   * Being hospitalized for a COPD exacerbation within the past year
   * Be using or be prescribed supplemental oxygen for 12 or more hours per day
   * Willingness to make return visits and availability by telephone for duration of study.

Exclusion Criteria:

1. A diagnosis of asthma established by each study investigator on the basis of the recent American Thoracic Society/European Respiratory Society and National Institute for Health and Care Excellence guidelines.
2. The presence of a diagnosis other than COPD that results in the patient being either medically unstable, or having a predicted life expectancy < 2 years.
3. Women who are at risk of becoming pregnant during the study (pre-menopausal) and who refuse to use acceptable birth control (hormone-based oral or barrier contraceptive) for the duration of the study.
4. Current tachy or brady arrhythmias requiring treatment
5. Presence of a pacemaker and/or internal cardioverter/defibrillator
6. Patients with a history of second or third degree (complete) heart block, or sick sinus syndrome
7. Baseline EKG revealing left bundle branch block, bifascicular block, ventricular tachyarrhythmia, atrial fibrillation, atrial flutter, supraventricular tachycardia (other than sinus tachycardia and multifocal atrial tachycardia), or heart block (2nd degree or complete)
8. Resting heart rate less than 65 beats per minute, or sustained resting tachycardia defined as heart rate greater than 120 beats per minute.
9. Resting systolic blood pressure of less than 100mm Hg.
10. Subjects with absolute (Class 1) indications for beta-blocker treatment as defined by the combined American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons Guidelines which include myocardial infarction, acute coronary syndrome, percutaneous coronary intervention or coronary artery bypass surgery within the prior 3 years and patients with known congestive heart failure defined as left ventricular ejection fraction <40%.(29, 30)
11. Critical ischemia related to peripheral arterial disease.
12. Other diseases that are known to be triggered by beta-blockers or beta-blocker withdrawal including myasthenia gravis, periodic hypokalemic paralysis, pheochromocytoma, and thyrotoxicosis
13. Patients on other cardiac medications known to cause atrioventricular (AV) node conduction delays such as amiodarone, digoxin, and calcium channel blockers including verapamil and diltiazem as well as patients taking clonidine.
14. Hospitalization for uncontrolled diabetes mellitus or hypoglycemia within the last 12 months.
15. Patients with cirrhosis
16. A clinical diagnosis of bronchiectasis defined as production of > one-half cup of purulent sputum/day.
17. Patients otherwise meeting the inclusion criteria will not be enrolled until they are a minimum of four weeks from their most recent acute exacerbation (i.e., they will not have received a course of systemic corticosteroids, an increased dose of chronically administered systemic corticosteroids, and/or antibiotics for an acute exacerbation for a minimum of four weeks).

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dransfield, MD, Principal Investigator — University of Alabama at Birmingham; John Connett, PhD, Principal Investigator — University of Minnesota; Stephen Lazarus, MD, Principal Investigator — University of California, San Francisco
Locations (27):
- United States (27):
  - Birmingham, Alabama VA Medical, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco-Fresno, Fresno, California
  - LA BioMed at Harbor-UCLA Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Louisiana State University, New Orleans, Louisiana
  - University of Maryland Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Veteran's Administration Medical Center, Minneapolis, Minnesota
  - HealthPartners Research Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian/Queens, Flushing, New York
  - Cornell University, Ithaca, New York
  - Columbia University, New York, New York
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - The University of Vermont, Burlington, Vermont
  - University of Washington School of Medicine, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parekh TM, Helgeson ES, Connett J, Voelker H, Ling SX, Lazarus SC, Bhatt SP, MacDonald DM, Mkorombindo T, Kunisaki KM, Fortis S, Kaminsky D, Dransfield MT. Lung Function and the Risk of Exacerbation in the beta-Blockers for the Prevention of Acute Exacerbations of Chronic Obstructive Pulmonary Disease Trial. Ann Am Thorac Soc. 2022 Oct;19(10):1642-1649. doi: 10.1513/AnnalsATS.202109-1042OC. PMID 35363600
- [Derived] Dransfield MT, Voelker H, Bhatt SP, Brenner K, Casaburi R, Come CE, Cooper JAD, Criner GJ, Curtis JL, Han MK, Hatipoglu U, Helgeson ES, Jain VV, Kalhan R, Kaminsky D, Kaner R, Kunisaki KM, Lambert AA, Lammi MR, Lindberg S, Make BJ, Martinez FJ, McEvoy C, Panos RJ, Reed RM, Scanlon PD, Sciurba FC, Smith A, Sriram PS, Stringer WW, Weingarten JA, Wells JM, Westfall E, Lazarus SC, Connett JE; BLOCK COPD Trial Group. Metoprolol for the Prevention of Acute Exacerbations of COPD. N Engl J Med. 2019 Dec 12;381(24):2304-2314. doi: 10.1056/NEJMoa1908142. Epub 2019 Oct 20. PMID 31633896
- [Derived] Bhatt SP, Connett JE, Voelker H, Lindberg SM, Westfall E, Wells JM, Lazarus SC, Criner GJ, Dransfield MT. beta-Blockers for the prevention of acute exacerbations of chronic obstructive pulmonary disease (betaLOCK COPD): a randomised controlled study protocol. BMJ Open. 2016 Jun 7;6(6):e012292. doi: 10.1136/bmjopen-2016-012292. PMID 27267111

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoprolol Succinate | Placebo
Started | 268 | 264
Completed | 268 | 264
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoprolol Succinate | Placebo | Total
Number analyzed (Participants) | 268 | 264 | 532
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 125 | 247
  >=65 years | 146 | 139 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (7.6) | 64.8 (7.9) | 65.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 123 | 247
  Male | 144 | 141 | 285
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 178 | 194 | 372
  Black | 83 | 60 | 143
  Other | 7 | 10 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 268 | 264 | 532
FEV1 after bronchodilation - % of predicted value [Mean (Standard Deviation); unit: % of predicted value] | 41.3 (16.3) | 40.8 (16.2) | 41.1 (16.3)
FEV1:FVC ratio - % [Mean (Standard Deviation); unit: ratio %] | 44.2 (11.7) | 45.2 (21.6) | 44.7 (17.3)
Smoking history No. of pack-yr [Mean (Standard Deviation); unit: pack-years] | 50.7 (28.7) | 49.5 (29.6) | 50.1 (29.1)
Systolic Blood pressure - mm Hg [Mean (Standard Deviation); unit: mm Hg] | 128.4 (16.5) | 130.6 (15.9) | 129.5 (16.2)
Diastolic Blood pressure - mm Hg [Mean (Standard Deviation); unit: mm Hg] | 77.2 (9.2) | 76.8 (9.1) | 77.0 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of an Acute COPS Exacerbation
Description: Acute exacerbations are defined as a "complex of respiratory symptoms (increase or new onset) of more than one of the following: cough, sputum, wheezing, dyspnea, or chest tightness requiring treatment with antibiotics and/or systemic steroids for at least three days".
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
days | 202 [162 to 282] | 222 [189 to 295]

2. Secondary Outcome: Number of Acute Exacerbations of COPD
Description: Number of acute exacerbations of COPD - rate per person-year
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: no. of events/person-yr
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
no. of events/person-yr | 1.40 [1.21 to 1.61] | 1.33 [1.15 to 1.54]

3. Secondary Outcome: Number of Emergency Department Visits Resulting From Acute Exacerbations of COPD
Description: Number of Emergency Department visits resulting from acute exacerbations of COPD - rate
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: events per person-year
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
events per person-year | 0.17 [0.11 to 0.25] | 0.18 [0.12 to 0.26]

4. Secondary Outcome: Number of Hospital Admissions Resulting From Acute Exacerbations of COPD
Description: Number of hospital admissions resulting from acute exacerbations of COPD - rate
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: events per person-year
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
events per person-year | 0.66 [0.47 to 0.86] | 0.42 [0.30 to 0.55]

5. Secondary Outcome: Hospital Days Resulting From Acute Exacerbations of COPD
Description: Number of hospital days resulting from acute exacerbations of COPD reported as negative binomial estimates of mean hospital days per patient year.
Time Frame: 14 months
Measure: Mean (95% Confidence Interval); unit: hospital days
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
hospital days | 3.09 [2.05 to 4.64] | 0.96 [0.62 to 1.48]

6. Secondary Outcome: Major Adverse Cardiovascular Events
Description: Major adverse cardiovascular events (MACE), percutaneous coronary intervention or coronary artery bypass grafting. MACE defined by cardiovascular death, hospitalization for myocardial infarction, heart failure, or stroke
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
Participants
  Myocardial Infarction | 2 | 1
  Heart Failure | 2 | 3
  Stroke | 1 | 1
  Sudden Cardiac Death | 0 | 1

7. Secondary Outcome: All-cause Mortality
Description: All-cause mortality count
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
Participants | 11 | 5

8. Secondary Outcome: Incidence of Presumed Metoprolol-related Side-effects
Description: New or worsened (Neural: depression, headache, syncope, seizures, somnolence, memory loss, loss of sexual desire or erectile dysfunction, and fatigue; Hypersensitivity: rash, pruritus, tongue or facial swelling; Gastrointestinal: diarrhea, vomiting, nausea or constipation; Cardiovascular: bradycardia and hypotension as discussed below; Respiratory: bronchospasm and changes in lung function as discussed below).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
Participants
  Depression | 28 | 39
  Headache | 71 | 78
  Fainting | 4 | 8
  Daytime Sleepiness | 58 | 70
  Memory Loss | 20 | 21
  Loss of sexual desire or erectile dysfunction | 10 | 6
  Lack of energy | 91 | 77
  Rash | 17 | 21
  Itching | 11 | 18
  Tongue or facial swelling | 7 | 5
  Vomiting | 11 | 18
  Nausea | 45 | 42
  Constipation | 30 | 32
  Wheezing | 88 | 79
  Shortness of breath | 115 | 112
  Chest tightness | 81 | 80
  Heart skipping or irregular beats | 16 | 15
  Dizziness/light headedness | 74 | 64

9. Secondary Outcome: Modified Medical Research Council Dyspnea Scale (MMRC)
Description: Modified Medical Research Council Dyspnea Scale (MMRC) change from baseline to visit day 336. The MMRC scale is a five-point scale originally published in 1959 that considers certain activities, such as walking or climbing stairs, which provoke breathlessness. Scale from 0 to 4 with lower scores indicating less breathlessness.
Time Frame: 1 year
Population: Participants with data at baseline and visit day 336
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 207 | 201
score on a scale | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]

10. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in FEV1 % Predicted from baseline to visit day 336 as assessed by spirometry
Time Frame: 1 year
Population: Participants with data at baseline and visit day 336
Measure: Mean (95% Confidence Interval); unit: percentage of predicted
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 193 | 197
percentage of predicted | -2.24 [-3.28 to -1.20] | -1.46 [-2.50 to -0.42]

11. Secondary Outcome: Exercise Capacity as Assessed by the 6 Minute Walk Distance (6MWD)
Description: 6MWD change from baseline to visit day 336. The 6MWD has been used as a simple tool to assess overall exercise tolerance in patients with chronic cardiopulmonary disease including COPD.
Time Frame: Baseline, 1 year
Population: Participants with data at baseline and visit day 336
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 174 | 166
meters | -17.64 [-28.75 to -6.53] | -11.87 [-23.21 to -0.54]

12. Secondary Outcome: Markers of Systemic Inflammation
Description: Fibrinogen: assessed at screening/randomization and at conclusion of the study to determine if beta-blockade impacts levels of systemic inflammation that portend overall cardiac risk.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
mg/dL
  Fibrinogen baseline | 384.8 (94.6) | 378.2 (91.9)
  Fibrinogen Visit 336 | 392.5 (90.5) | 386.0 (110.0)

13. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ)
Description: SGRQ change from baseline to visit day 336. The SGRQ total score change from baseline. SGRQ is a respiratory specific health status questionnaire with scores ranging from 0 to 100. The lower score indicates a better health status.
Time Frame: Baseline, 1 year
Population: Participants with data at baseline and visit day 336
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 203 | 200
score on a scale | 0.52 [-1.01 to 2.04] | -0.25 [-1.79 to 1.28]

14. Secondary Outcome: COPD Assessment Test (CAT)
Description: COPD Assessment Test (CAT) change from baseline. The CAT is a simple, eight item, health status instrument for patients with COPD that provides a score of 0-40. Lower scores denote better health status.
Time Frame: Baseline, 1 year
Population: Participants with data at baseline and visit day 336
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 206 | 200
score on a scale | 0.88 [0.07 to 1.69] | -0.59 [-1.41 to 0.23]

15. Secondary Outcome: San Diego Shortness of Breath Questionnaire (SOBQ)
Description: San Diego Shortness of Breath Questionnaire (SOBQ) change from baseline. A 24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living. Each item has a 6-point scale (0 = "not at all" to 5 = "maximal or unable to do because of breathlessness").
Time Frame: 1 year
Population: Participants with data at baseline and visit day 336
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 204 | 199
score on a scale | 0.52 [-1.01 to 2.04] | -0.25 [-1.79 to 1.28]

16. Secondary Outcome: Acute Exacerbations of COPD and MACE
Description: MACE defined by cardiovascular death, hospitalization for myocardial infarction, heart failure, or stroke
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 268 | 264
Participants
  Myocardial Infarction | 2 | 1
  Heart Failure | 2 | 3
  Stroke | 1 | 1
  Sudden cardiac death | 0 | 1
  COPD Exacerbation (Serious) | 55 | 32

17. Secondary Outcome: Short Form Health Survey (SF-36) Physical Function Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. 8 multi-item scales with higher score indicating better health state. The Physical Functioning scale is 10 items assessing the extent to which health limits physical activities such as self-care, walking, climbing stairs, bending lifting, and moderate and vigorous activities transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 30.0 [15.0 to 50.0] | 30.0 [15.0 to 45.0]
  Day 112 visit | 30.0 [15.0 to 55.0] | 30.0 [15.0 to 50.0]
  Day 336 Visit | 30.0 [15.0 to 50.0] | 35.0 [15.0 to 50.0]

18. Secondary Outcome: Short Form Health Survey (SF-36) Role Functioning - Physical Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. Includes 8 multi-item scales with higher score indicating better health state. The Role Functioning - Physical Scale contains 4 items assessing the extent to which physical health interferes with work or other daily activities, including accomplished less than wanted, limitations in the kind of activities. Items are transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 25.0 [0.0 to 50.0] | 25.0 [0.0 to 56.2]
  Day 112 visit | 25.0 [0.0 to 75.0] | 25.0 [0.0 to 75.0]
  Day 336 Visit | 12.5 [0.0 to 75.0] | 12.5 [0.0 to 50.0]

19. Secondary Outcome: Short Form Health Survey (SF-36) Role Functioning - Emotional Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. Includes 8 multi-item scales with higher score indicating better health state. The Role Functioning - Emotional Scale includes 3 items assessing extent to which emotional problems interfere with work or other daily activities. Items are transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 100.0 [0.0 to 100.0] | 66.7 [0.0 to 100.0]
  Day 112 visit | 66.7 [0.0 to 100.0] | 66.7 [0.0 to 100.0]
  Day 336 Visit | 66.7 [0.0 to 100.0] | 66.7 [0.0 to 100.0]

20. Secondary Outcome: Short Form Health Survey (SF-36) Energy/Fatigue Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. Includes 8 multi-item scales with higher score indicating better health state. The Energy/Fatigue Scale includes 4 items. Items are transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 50.0 [35.0 to 60.0] | 50.0 [35.0 to 60.0]
  Day 112 visit | 50.0 [35.0 to 60.0] | 45.0 [30.0 to 60.0]
  Day 336 Visit | 50.0 [35.0 to 60.0] | 45.0 [30.0 to 55.0]

21. Secondary Outcome: Short Form Health Survey (SF-36) Emotional Well-being Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. Includes 8 multi-item scales with higher score indicating better health state. The Emotional Well-being Scale includes 5 items assessing emotional wellbeing. Items are transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 76.0 [60.0 to 84.0] | 72.0 [56.0 to 84.0]
  Day 112 visit | 76.0 [60.0 to 88.0] | 72.0 [56.0 to 84.0]
  Day 336 Visit | 76.0 [60.0 to 88.0] | 72.0 [56.0 to 84.0]

22. Secondary Outcome: Short Form Health Survey (SF-36) Social Functioning Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. Includes 8 multi-item scales with higher score indicating better health state. The Social Functioning Scale includes 2 items assessing extent to which physical health or emotional problems interfere with normal social activities. Items are transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 62.5 [50.0 to 87.5] | 62.5 [50.0 to 87.5]
  Day 112 visit | 62.5 [50.0 to 87.5] | 62.5 [50.0 to 87.5]
  Day 336 Visit | 75.0 [50.0 to 87.5] | 62.5 [37.5 to 87.5]

23. Secondary Outcome: Short Form Health Survey (SF-36) Bodily Pain Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. Includes 8 multi-item scales with higher score indicating better health state. The Bodily Pain Scale includes 2 items assessing the intensity of pain and effect of pain on normal work, both inside and outside the house. Items are transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 67.5 [45.0 to 90.0] | 67.5 [45.0 to 90.0]
  Day 112 visit | 67.5 [45.0 to 90.0] | 67.5 [45.0 to 90.0]
  Day 336 Visit | 57.5 [35.0 to 90.0] | 57.5 [42.5 to 87.5]

24. Secondary Outcome: Short Form Health Survey (SF-36) General Health Scale
Description: Short Form Health Survey (SF-36) is a generic tool to assess overall health status and allows comparison between different diseases. Includes 8 multi-item scales with higher score indicating better health state. The General Health Scale includes 4 items assessing personal evaluations of health. Items are transformed to a score with a range of 0-100.
Time Frame: 1 year
Population: Participants with SF-36 data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Metoprolol Succinate | Placebo
Number analyzed (Participants) | 265 | 262
Units on a scale
  Baseline | 40.0 [25.0 to 55.0] | 40.0 [25.0 to 55.0]
  Day 112 visit | 40.0 [25.0 to 55.0] | 35.0 [25.0 to 55.0]
  Day 336 Visit | 40.0 [25.0 to 55.0] | 35.0 [25.0 to 50.0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Metoprolol Succinate | Placebo
All-Cause Mortality (participants affected / at risk) | 11/268 | 5/264
Serious Adverse Events (participants affected / at risk) | 86/268 | 59/264
Other Adverse Events (participants affected / at risk) | 162/268 | 157/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoprolol Succinate (N=268) | Placebo (N=264)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2) | 3 (3)
Stroke (Cardiac disorders) | 1 (1) | 1 (2)
Arrhythmias (Cardiac disorders) | 2 (2) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Other Cardiovascular (Cardiac disorders) | 1 (1) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 55 (72) | 32 (47)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 11 (12)
Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 2 (3) | 5 (5)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Other Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Infections, non-pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Head, eyes, ears, nose and throat (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Trauma/Falls (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Neurologic, non-stroke (Nervous system disorders) | 1 (1) | 1 (1)
Psychiatric (Psychiatric disorders) | 1 (1) | 0 (0)
Chest Pain, not otherwise specified (Cardiac disorders) | 1 (1) | 1
Endocrine (Endocrine disorders) | 1 (1) | 0 (0)
Other (General disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoprolol Succinate (N=268) | Placebo (N=264)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 115 (205) | 122 (209)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 19 (24)
Acute Sinusitis (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 10 (12)
Headache (General disorders) | 18 (21) | 15 (16)
Gastrointestinal symptoms (Gastrointestinal disorders) | 24 (29) | 30 (36)
Dizziness (General disorders) | 23 (27) | 16 (17)
Respiratory Infections (Infections and infestations) | 30 (34) | 23 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02587351/Prot_SAP_000.pdf